CLINICAL TRIAL: NCT02021851
Title: THE EFFECT OF THE COMBINATION OF DEXAMETHASONE WITH ONDANSETRON VERSUS DEXAMETHASONE WITH APREPITANT TO PREVENT POSTOPERATIVE NAUSEA AND VOMITING IN PATIENTS UNDERGOING LAPAROSCOPIC SURGERY
Brief Title: Prevention of Nausea and Vomiting in Patients After Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Sevgi Bilgen, Assistant professor, Yeditepe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 125
Record Dates: First submitted 2013-12-09; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Dexamethasone,; Ondansetron; Aprepitant; PONV; Laparoscopic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Aprepitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group DA: Dexamethasone and aprepitant (Active Comparator): Group DA: Dexamethasone: 8 mg (intravenous), Aprepitant: 40 mg (oral)
  Interventions: Drug: Dexamethasone and aprepitant
- Group DO: Dexamethasone and ondansetron (Placebo Comparator): Group DO: Dexamethasone: 8 mg (intravenous), Ondansetron: 4 mg (intravenous)
  Interventions: Drug: Dexamethasone and ondansetron

INTERVENTIONS:
Drug: Dexamethasone and aprepitant
  Arms: Group DA: Dexamethasone and aprepitant
Drug: Dexamethasone and ondansetron
  Arms: Group DO: Dexamethasone and ondansetron

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common problem after general anesthesia. The incidence can be as high as 80 percent in high-risk patients. Investigators designed this randomized, double- blind, single-center study to compare the efficacy of the combination of dexamethasone with ondansetron and dexamethasone with aprepitant undergoing laparoscopic surgery.

Seventy American Society of Anesthesiologist (ASA) physical class I-II, age 18-60 years patients scheduled for laparoscopic surgery were included in this study. Anesthesia was induced with propofol, fentanyl, and rocuronium, and maintained with sevoflurane in oxygen / air mixture in all patients. Remifentanil was continuously infused during surgery. Patients were randomly divided into two groups. Patients in the dexamethasone and aprepitant group (group DA, n=35) received 40 mg aprepitant orally 1 to 2 hours before induction of anesthesia and 2 ml saline intravenous (iv) within the last 30 minutes of surgery. Patients in the dexamethasone and ondansetron group (group DO, n=35) received an oral placebo identical to aprepitant 1 to 2 hours before induction of anesthesia and 4 mg ondansetron iv within the last 30 minutes of surgery. All patient received iv 8 mg dexamethasone after induction of anesthesia.

PONV and postoperative opioid consumption were assessed for 24 hours postoperatively. The blindly evaluated primary outcome was complete response. The secondary outcomes were incidence of nausea, retching or vomiting, the need of rescue antiemetic and opioid consumption within 24 hours after surgery. Statistical analyses were performed using Mann-Whitney U test, Chi-square test, and Fisher's Exact test. P<0.05 was considered statistically significant.Investigators hypothesized that the antiemetic efficacy of the aprepitant and dexamethasone combination is superior compared with ondansetron and dexamethasone combination following the laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 60 Years
* ASA (American Society of Anesthesiologist) physical status I or II
* Patients undergoing laparoscopic gynecologic surgery or laparoscopic cholecystectomy

Exclusion Criteria:

* Hypersensitivity or contraindication to the study medications,
* Antiemetic drug or steroid use within 24 hours before anesthesia,
* History of diabetes mellitus,
* History of motion sickness or postoperative nausea and vomiting,
* Pregnancy,
* Breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Complete response | One year
  The primary outcome is complete response: A complete response is defined as no postoperative nausea (VRS≤3), retching or vomiting and no need for rescue antiemetic.

SECONDARY OUTCOMES:
Nausea | One year
  The secondary outcome measure is incidence of nausea
Retching | One year
  The secondary outcome measure is incidence of retching
Vomiting | One year
  The secondary outcome measure is incidence of vomiting
Need of rescue antiemetic | One year
  The secondary outcome measure is incidence of the need of rescue antiemetic within 24 hours after surgery.

OTHER OUTCOMES:
Opioid consumption | One year
  Opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Hospital, Devlet Yolu, Ankara Cad 102/104, Kozyatagi Istanbul, Turkey (Türkiye)